CLINICAL TRIAL: NCT05257785
Title: Lymfit to Improve the Fitness and Quality of Life in Lymphoma Survivors: A Randomized Controlled Trial
Brief Title: Lymfit to Improve the Fitness and Quality of Life in Lymphoma Survivors
Acronym: Lymfit_RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Jewish General Hospital (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Christine Maheu, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-2560
Record Dates: First submitted 2022-02-09; First posted 2022-02-25 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Lymphoma; Cancer Survivors
Keywords: Cancer survivorship; Quality of Life; Physical Activity; Fear of Recurrence; Randomized controlled trial
MeSH Terms: conditions — Lymphoma; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymfit exercise intervention (Experimental): Participants randomized to the intervention group will be allocated a pre-registered Fitbit, a personalized exercise prescription designed by the kinesiologist, and 12 weeks of supervision by the kinesiologist.
  Interventions: Behavioral: Lymfit exercise intervention
- Waitlist control (Other): Participants will receive the exact same Lymfit exercise intervention 3 months after they consent to participate in the study.
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Lymfit exercise intervention — Participants randomized to this arm will be allocated a pre-registered Inspire II / Charge IV model Fitbit. The kinesiologist of the study will meet with the participants for a baseline fitness assessment. The kinesiologist will examine the baseline physical activity levels, fitness level and sedentary behaviours of the participants, to design a personalized exercise prescription. Within one week after the baseline fitness assessment, the kinesiologist will contact the participants to discuss the exercise prescription. Every two weeks there-after, the kinesiologist will follow up with the participants via videoconferencing to discuss their progress and to modify or advance their exercise prescriptions as needed. Participants will be followed-up at 6 months and 12 months.
  Arms: Lymfit exercise intervention
Behavioral: Waitlist control — Participants will be contacted by the study kinesiologist for a baseline fitness assessment 3 months after they consent, participants will be given a Fitbit, a personalized exercise prescription and receive bi-weekly follow-ups for 12 weeks.
  Arms: Waitlist control

SUMMARY:
This randomized control trial seeks to determine whether a tailored and supervised exercise program adopting mobile-health technology will be able to improve fitness and quality of life among lymphoma survivors.

DETAILED DESCRIPTION:
Lymphoma is the most common cancer diagnosed in young adults. While curing 80% of patients, lymphoma treatment has a significant impact on young adults' health and psycho-social wellbeing by increasing fatigue and anxiety, risk of cardiovascular disease and other chronic disorders, all of which compromise one's quality of life. Regular exercise has the potential to reduce the side effects associated with cancer treatments. Thus, the most recent guidelines suggest that cancer patients should engage in adapted exercise programs during and after their treatment.

However, these guidelines are not systematically recommended by doctors and are often not followed by patients. Fatigue and lack of motivation are the main barriers to exercise among cancer survivors. Our study aims to identify young adults lymphoma patients and encourage them to adhere to the exercise guidelines with the help of an exercise physiologist and a fitness tracker. The investigators will evaluate the efficacy of these strategies in motivating exercise among young adults lymphoma survivors. Our proposed study carries significant implications for the prevention of complications of treatment for young adults lymphoma survivors.

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed lymphoma patients who received an initial diagnosis at the age of age 18-39,
2. approved by their hematologist as having no contra-indications to vigorous exercise,
3. receiving or has received chemotherapy with curative intent within the past 6 months,
4. own a cellular phone that is able to download the Fitbit app and to complete the study questionnaires online in either French or English, and
5. has an Internet connection at home that supports participation in coaching sessions via videoconferencing (zoom).

Exclusion Criteria:

1. The patient has contra-indications to vigorous exercise,
2. the patient doesn't want to wear a fitness tracker due to various concerns (as no Fitbit data could be collected).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of the exercise guideline as determined by comparing the active minutes captured in the Fitbit | 3 months
  The investigators will determine the percentage of lymphoma patients who adhere to the recommended exercise guidelines for cancer patients at baseline and after the intervention, i.e. compare the minutes of Moderate to vigorous physical activity per week captured in the Fitbit among participants in the intervention arm and waitlist control arm at baseline and 3 months.

SECONDARY OUTCOMES:
Change from baseline multi-dimensional Quality of life (QoL) assessed by the Patient-Reported Outcomes Measurement Information System-29 | 12 months
  The Patient-Reported Outcomes Measurement Information System-29 is a 29-item instrument assessing multi-dimensional eight domains (29 items) (i.e., anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, ability to participate in social roles and activities, and pain intensity). Raw scores generated for each domain are transformed into T scores; higher T scores indicate greater endorsement of the construct being assessed.
Change from baseline Work Ability assessed by the Work Ability Index (WAI) | 12 months
  The Work Ability Index (WAI) questionnaire (7 items) will be used to collect productivity loss data within clinical trials and is suitable for direct translation into a monetary figure. The WAI measured in this way ranges from 7 to 49 points and 4 categories have been suggested to describe WAI levels: poor [7-27], moderate [28-36], good (37-43) and excellent (44-49).
Change from baseline Fear of Cancer Recurrence assessed by the Cancer Worry Scale (CWS) | 12 months
  Cancer Worry Scale is a six-item scale designed to measure worry about the risk of developing cancer and the impact of worry on daily functioning. The scale consists of six questions with four response options (1 = not at all or rarely; 2 = sometimes; 3 = often; 4 = almost all the time), such that each individual attains a score ranging from 6 (minimum worry) to 24 (maximum worry).

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided